CLINICAL TRIAL: NCT05032144
Title: A Randomized,Double-blind,Placebo-controlled,Single-ascending Dose Phase Ⅰa Study to Evaluate the Safety,Tolerability,Pharmacokinetics and Pharmacodynamics of STSA-1002 Following Intravenous Infusion in Healthy Subjects
Brief Title: The Safety and Tolerability of STSA-1002 Following Intravenous Infusion in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSA-1002-01
Record Dates: First submitted 2021-08-19; First posted 2021-09-02 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2021-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1:2mg/kg (Experimental): All participants (fasted) received either 2mg/kg of STSA-1002 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1002 injection; Drug: Placebo
- Cohort 2:5mg/kg (Experimental): All participants (fasted) received either 5mg/kg of STSA-1002 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1002 injection; Drug: Placebo
- Cohort 3:10mg/kg (Experimental): All participants (fasted) received either 10mg/kg of STSA-1002 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1002 injection; Drug: Placebo
- Cohort 4:20mg/kg (Experimental): All participants (fasted) received either 20mg/kg of STSA-1002 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1002 injection; Drug: Placebo
- Cohort 5:30mg/kg (Experimental): All participants (fasted) received either 30mg/kg of STSA-1002 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1002 injection; Drug: Placebo

INTERVENTIONS:
Drug: STSA-1002 injection — Intravenous injection
  Arms: Cohort 1:2mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 1:2mg/kg
Drug: STSA-1002 injection — Intravenous injection
  Arms: Cohort 2:5mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 2:5mg/kg
Drug: STSA-1002 injection — Intravenous injection
  Arms: Cohort 3:10mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 3:10mg/kg
Drug: STSA-1002 injection — Intravenous injection
  Arms: Cohort 4:20mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 4:20mg/kg
Drug: STSA-1002 injection — Intravenous injection
  Arms: Cohort 5:30mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 5:30mg/kg

SUMMARY:
A randomized,double-blind,placebo-controlled,single-ascending dose phase Ⅰa study to evaluate the safety,tolerability,pharmacokinetics and pharmacodynamics of STSA-1002 following intravenous infusion in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects,aged ≥18 but ≤65，male and female.
* Body mass index:18.0～32.0kg/m²，inclusive.
* Subjects(including their partners) agree to take highly effective contraceptive measures during the study,and they have no birth plan or sperm donation plan within 3months after the end of the study.
* Female and/or male subjects those meet the below criteria:

If a female subject of child bearing potential-agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the administration of IMP,during the study,and for at least 3 months after the end of the study. An acceptable method of contraception includes one of the following:

Abstinence from heterosexual intercourse Hormonal contraceptives(brith control pills,injectable/implant/insertable hormonal birth control products, transdermal patch) Intrauterine device(with or without hormones) OR agrees to use a double barrier method (e.g. condom and spermicide) . If a female subject of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in a menopausal state (at least 1 year without menses), as confirmed by Follicle-stimulating hormone (FSH) levels (≥ 40 mIU/mL).

A male subject that engages in sexual activity that has the risk of pregnancy must agree to use a double barrier method (e.g. condom and spermicide) and agree to not donate sperm during the study and for at least 3 months after the end of the study.

* Medical histories, physical examinations, laboratory examinations and study-related examinations and tests of the subjects show normal results or mild abnormalities with no clinical significance before enrollment, and the Investigator judges that they are eligible.
* Subjects are aware of the risks of the study, and voluntarily participate in the clinical study and sign an informed consent form (ICF).

Exclusion Criteria:

* History of cardiovascular, respiratory, kidney, liver, metabolism, endocrine, gastrointestinal, blood, nerve, skin and mental illness, cancer or other major disease that in the judgment of the Investigator might put the subject as risk on this study.
* History of tuberculosis or a recent history of infection within the past 4 weeks.
* History of recurrent infections.
* Presence of clinically significant laboratory values during the screening period, as defined by an Investigator.
* Presence of clinically significant vital signs values or of electrocardiogram (ECG) abnormalities during the screening period, as defined by an Investigator.
* Subjects who have autoimmune disease or immunodeficiency, or have a family history of related diseases.
* Subjects who have allergies, or have or are currently suffering from clinically significant atopic allergies, hypersensitivity or allergic reactions, including known or suspected clinically relevant hypersensitivity or allergic reactions to certain components of the IMP preparation, or a history of allergies to other drugs or biological agents.
* Positive screening test results for human immunodeficiency virus (HIV-1/HIV-2) antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCVAb).
* Subjects who have received treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to screening or 90 days for biologic compounds prior to screening.
* Subjects who have participated in any vaccine clinical study as subjects within 3 months before enrollment or plan to receive live vaccines during the study period, and subjects who have received vaccines 28 days prior to the IMP administration or plan to receive vaccines within 2 months after the end of the study.
* Subjects who have taken drugs that may affect immune function within 6 months before screening, have received any monoclonal antibody or biological agent for treatment (for any illness) within the previous 3 months, and have previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 7 days prior to IMP administration.
* Subjects whose daily consumption of coffee, tea and/or cola is more than 750 mL or 25 fl. oz in the last 30 days before enrollment.
* Subjects who have a positive urine alcohol test or urine drug test before enrollment.
* Subjects who have nicotine consumption (e.g., smoking, nicotine patch, nicotine chewing gum, or electronic cigarettes) within 3 months prior to screening and inability to refrain from nicotine consumption from screening until end of study.
* Female subjects who are pregnant or breastfeeding during the screening period and on admission.
* Subjects whose daily consumption of alcohol at the time of screening or at any time within the prior 6 months is more than 2 standard drinks, where 1 standard drink = 355 mL or 12 oz (1 can) of regular-strength (5%) beer; 150 mL or 5 oz wine; 45 mL or 1.5 oz liquor/spirits (40%).
* History of substance use disorder (within 1 year of screening).
* Subjects who have undergone major surgery within 2 months of screening, or who will have elective surgery that will occur during the study period.
* Subjects who have donated either more than approximately 500 mL of blood (exclusive plasma donation) within 56 days (8 weeks) prior to screening or any plasma within 7 days (1 week) prior to screening.
* Subjects fails or is unwilling to abstain from strenuous physical activities for at least 48 hours prior to IP administration and throughout the study.
* Subjects with any factors that would, in the Investigator's judgment, preclude them from participating in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Clinically Significant Laboratory Abnormalities,Clinically Significant Electrocardiogram Abnormalities, Clinically Significant Vital Signs Abnormalities And Clinically Significant Physical Examination Abnormalities | Day 1 through Day 51
Maximum plasma concentration(Cmax) | Up to 1200 hours postdose
Area under the plasma concentration-time curve from time 0 to the collection time point of the last measurable concentration(AUC 0-t) | Up to 1200 hours postdose
Area under the plasma concentration-time curve from time 0 to infinity(AUC0-∞) | Up to 1200 hours postdose
Time of maximum concentration(Tmax) | Up to 1200 hours postdose
Elimination half-life(t1/2) | Up to 1200 hours postdose
Elimination rate constant of plasma drug concentration in terminal phase(λz) | Up to 1200 hours postdose
Last measurable concentration(Clast) | Up to 1200 hours postdose
Mean residence time(MRT) | Up to 1200 hours postdose
Clearance(CL) | Up to 1200 hours postdose
Apparent volume of distribution(Vz) | Up to 1200 hours postdose

SECONDARY OUTCOMES:
Change from baseline in concentration of free C5a and anti-drug antibody | Up to 1200 hours postdose
  To evaluate the pharmacodynamics (PD) characteristics and immunogenicity of STSA-1002 in healthy subjects
Change from baseline in concentration of CH50,IL-6,IL-8,TNF-α,IFN-γ | Up to 1200 hours postdose
  To evaluate the effect of STSA-1002 on CH50, IL-6, IL-8, TNF-α, IFN-γ

CONTACTS AND LOCATIONS:
Locations (1):
- AltaSciences Clinical Kansas, Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No